CLINICAL TRIAL: NCT04831567
Title: Phase II Study of MIBG-I131 (Metaiodobenzylguanidine) in Patients With Well Differentiated Neuroendocrine Tumors and MIBG Positive Scan
Brief Title: Study of MIBG-I131 in Patients With Well Differentiated Neuroendocrine Tumors
Acronym: MIBNET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Rachel Riechelmann, Head of Medical Oncology Department, AC Camargo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3025/20
Record Dates: First submitted 2021-03-25; First posted 2021-04-05 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Neuroendocrine Tumors
Keywords: MIBG-I131; Nuclear medicine; Treatment
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Intervention Model Description: This is a single-arm, unicentric, single-stage, phase 2 clinical study of therapeutic metaiodobenzylguanidine (MIBG) for patients with metastatic well-differentiated neuroendocrine tumors and radiological progression or intolerance after standard lines of treatment and with MIBG positive scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional (Experimental): The participants will be submitted to metaiodobenzylguanidine 4 doses of 7.400 Mbq (million of Becquerels) (200 mCi). Each dose will be repeated with a minimum interval of 60 days.
  Interventions: Radiation: MIBG-I131

INTERVENTIONS:
Radiation: MIBG-I131 — Radiopharmaceutical

SUMMARY:
This is a single-arm, unicentric, single-stage, phase 2 clinical study of therapeutic metaiodobenzylguanidine (MIBG) for patients with metastatic well-differentiated neuroendocrine tumors and radiological progression or intolerance after standard lines of treatment and with MIBG positive scan.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NET) are rare neoplasms, which frequently present metastatic and incurable at diagnosis. In this context, few effective therapies exist. When the disease becomes refractory to standard therapies, treatments with limited efficacy (eg, surgical debulking, cytotoxic chemotherapies, interferon alpha) that could lead to important adverse events are used. Therefore, clinical studies that test new therapeutic strategies in NET patients with refractory disease are needed. Treatment with radiopharmaceuticals have been studied in NET and showed to be promisor. As an example, is the treatment with Lutetium177 octreotate, disponible in Brazil for decades, and one of the most active therapeutic options to NET.

The radiopharmaceutical MIBG-I131 (metaiodobenzylguanidine linked to Iodine131) is the first treatment choice for patients with paraganglioma/pheochromocytoma (PggF), a rare type of neuroendocrine neoplasm originated from neural ganglia. Patients with this neoplasia are submitted to scintigraphy with MIBG-I131, a norepinephrine analog whose transporter protein is highly expressed in this tumor. If the uptake is positive, patients receive treatment with therapeutic doses of MIBG-I131. The disease control with this intervention could last two years. Old and small studies suggested that MIBG-I131 could also have an activity in other NET besides PggF. Gastrointestinal (GI) or lung NET could have a positive expression on MIBG-I131 scan in up to 50% of the cases. With this rationale, retrospective series reported that MIBG-I131 could offer clinical benefit in patients with GI NET, with disease control in up to 80% of the cases. However, the literature regarding therapeutic MIBG-I131 to NET not PggF is scarce, heterogeneous regarding population, methods of response assessment, doses of the radiopharmaceutical, and short follow-up time. Therefore, due to the absence of effective therapeutic options for patients with metastatic well-differentiated NET refractory to standard treatments, the evidence that NET can have a positive expression on MIBG-I131 scan, and that small retrospective studies with a low level of evidence suggest a benefit for control disease and improvement of symptoms, the investigators proposed a phase II study of MIBG-I131 to well-differentiated GI or lung NET patients with positive MIBG-I131 scan.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Histological diagnosis of well-differentiated neuroendocrine tumor (NET) (typical and atypical lung carcinoids and NET of all gastroenteropancreatic sites according to World Health Organization (WHO) 2019 classification); metastatic/unresectable, with no possibility of curative treatment.
* MIBG-I131 positive scan in at least one lesion with uptake compatible with therapeutic effectiveness.
* Disease with radiological progression (at least 10 percent tumor volume growth) in the last 12 months before day 1 cycle 1.
* Intolerance due to toxicities or lack of access to standard treatments - [private context (somatostatin analog, everolimus) and public health system (somatostatin analog)].
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance scale 0 to 2.
* Adequate organic function as defined by the following criteria:

  * serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal of the local laboratory (ULN-LL);
  * Total serum bilirubin ≤ 2.0 x ULN-LL;
  * Absolute neutrophil count ≥ 1,500 / mm^3;
  * Platelet count ≥ 100,000 / mm^3;
  * Hemoglobin ≥ 9.0 g / dL;
  * Estimated creatinine clearance by the Modification of Diet in Renal Disease (MDRD) equation ≥ 60ml / min
* Term of free and informed consent signed by the patient or legal representative.

Exclusion Criteria:

* Patients already treated with MIBG-I131.
* A history of serious clinical or psychiatric illness that, by clinical judgment, may involve participation risk in this study.
* Patients participating in other protocols with experimental drugs.
* Patients who underwent major recent surgery less than 4 weeks previously.
* Patients receiving chemotherapy or other oncologic therapy for less than 3 weeks.
* Pregnant or lactating patients.
* Another synchronous neoplasm that requires systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) at 6 months after the end of treatment | At 6 months after the end of MIBG-I131 (4 cycles - each cycle is 60 days)
  Defined by absence of radiological progression in conventional imaging examinations by RECIST 1.1.
Quality of life measured by questionnaire | At 6 months after the end of MIBG-I131 (4 cycles - each cycle is 60 days)
  Quality of life questionnaire (QLQ), assessed by the European Organisation for Research and Treatment of Cancer Quality of Life for Neuroendocrine Tumors (EORTC QLQ-GINET21) (score ranging from 0 to 100, with higher scores meaning better state of the patient). Improvement in at least 10% of the baseline score will be considered positive.

SECONDARY OUTCOMES:
Disease control rate (DCR) at 3 months after the end of treatment | At 3 months after the end of MIBG-I131 (4 cycles - each cycle is 60 days)
  Defined by absence of radiological progression in conventional imaging examinations by RECIST 1.1.
Progression-free survival | Trough study completion, an average of 3 years
  Defined by time from day 1 cycle 1 to death from any cause or radiological progression by RECIST 1.1, whichever occurs first. Patients alive and without progression at the time of study analysis will be censored for time-to-event analysis.
Radiological response rate | Trough study completion, an average of 3 years
  Assessed by RECIST 1.1 criteria.
Rate of Biochemical response | Trough study completion, an average of 3 years
  Defined by at least 30 percent drop in the tumor marker (24-hour urine 5-hydroxyindoleacetic acid (5-HIAA) and/or specific hormone), if functioning syndrome, at any time of treatment in relation to pre-treatment value.
Quality of life measured by questionnaires | Trough study completion, an average of 3 years
  Quality of life questionnaire (QLQ), assessed by the European Organisation for Research and Treatment of Cancer Quality of Life for Neuroendocrine Tumors (EORTC QLQ-GINET21) (score ranging from 0 to 100, with higher scores meaning better state of the patient). Improvement in at least 10% of the baseline score will be considered positive.
Incidence of Treatment-related Adverse Events assessed by Common Terminology Criteria for Adverse Events (CTCAE) | Trough study completion, an average of 3 years
  Frequency of adverse events of grades 2 or more by CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel SP Riechelmann, Phd, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057
- [Background] Strosberg J, El-Haddad G, Wolin E, Hendifar A, Yao J, Chasen B, Mittra E, Kunz PL, Kulke MH, Jacene H, Bushnell D, O'Dorisio TM, Baum RP, Kulkarni HR, Caplin M, Lebtahi R, Hobday T, Delpassand E, Van Cutsem E, Benson A, Srirajaskanthan R, Pavel M, Mora J, Berlin J, Grande E, Reed N, Seregni E, Oberg K, Lopera Sierra M, Santoro P, Thevenet T, Erion JL, Ruszniewski P, Kwekkeboom D, Krenning E; NETTER-1 Trial Investigators. Phase 3 Trial of 177Lu-Dotatate for Midgut Neuroendocrine Tumors. N Engl J Med. 2017 Jan 12;376(2):125-135. doi: 10.1056/NEJMoa1607427. PMID 28076709
- [Background] Riechelmann RP, Weschenfelder RF, Costa FP, Andrade AC, Osvaldt AB, Quidute AR, Dos Santos A, Hoff AA, Gumz B, Buchpiguel C, Vilhena Pereira BS, Lourenco Junior DM, da Rocha Filho DR, Fonseca EA, Riello Mello EL, Makdissi FF, Waechter FL, Carnevale FC, Coura-Filho GB, de Paulo GA, Girotto GC, Neto JE, Glasberg J, Casali-da-Rocha JC, Rego JF, de Meirelles LR, Hajjar L, Menezes M, Bronstein MD, Sapienza MT, Fragoso MC, Pereira MA, Barros M, Forones NM, do Amaral PC, de Medeiros RS, Araujo RL, Bezerra RO, Peixoto RD, Aguiar S Jr, Ribeiro U Jr, Pfiffer T, Hoff PM, Coutinho AK. Guidelines for the management of neuroendocrine tumours by the Brazilian gastrointestinal tumour group. Ecancermedicalscience. 2017 Jan 26;11:716. doi: 10.3332/ecancer.2017.716. eCollection 2017. PMID 28194228
- [Background] van Hulsteijn LT, Niemeijer ND, Dekkers OM, Corssmit EP. (131)I-MIBG therapy for malignant paraganglioma and phaeochromocytoma: systematic review and meta-analysis. Clin Endocrinol (Oxf). 2014 Apr;80(4):487-501. doi: 10.1111/cen.12341. Epub 2013 Nov 19. PMID 24118038
- [Background] Ezziddin S, Logvinski T, Yong-Hing C, Ahmadzadehfar H, Fischer HP, Palmedo H, Bucerius J, Reinhardt MJ, Biersack HJ. Factors predicting tracer uptake in somatostatin receptor and MIBG scintigraphy of metastatic gastroenteropancreatic neuroendocrine tumors. J Nucl Med. 2006 Feb;47(2):223-33. PMID 16455627
- [Background] Riechelmann RP, Pereira AA, Rego JF, Costa FP. Refractory carcinoid syndrome: a review of treatment options. Ther Adv Med Oncol. 2017 Feb;9(2):127-137. doi: 10.1177/1758834016675803. Epub 2016 Nov 2. PMID 28203303
- [Background] Kane A, Thorpe MP, Morse MA, Howard BA, Oldan JD, Zhu J, Wong TZ, Petry NA, Reiman R Jr, Borges-Neto S. Predictors of Survival in 211 Patients with Stage IV Pulmonary and Gastroenteropancreatic MIBG-Positive Neuroendocrine Tumors Treated with 131I-MIBG. J Nucl Med. 2018 Nov;59(11):1708-1713. doi: 10.2967/jnumed.117.202150. Epub 2018 May 18. PMID 29777005
- [Background] Mulholland N, Chakravartty R, Devlin L, Kalogianni E, Corcoran B, Vivian G. Long-term outcomes of (131)Iodine mIBG therapy in metastatic gastrointestinal pancreatic neuroendocrine tumours: single administration predicts non-responders. Eur J Nucl Med Mol Imaging. 2015 Dec;42(13):2002-12. doi: 10.1007/s00259-015-3116-4. Epub 2015 Jul 5. PMID 26142730
- [Background] Navalkissoor S, Alhashimi DM, Quigley AM, Caplin ME, Buscombe JR. Efficacy of using a standard activity of (131)I-MIBG therapy in patients with disseminated neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2010 May;37(5):904-12. doi: 10.1007/s00259-009-1326-3. Epub 2009 Dec 17. PMID 20016892
- [Background] Bomanji JB, Wong W, Gaze MN, Cassoni A, Waddington W, Solano J, Ell PJ. Treatment of neuroendocrine tumours in adults with 131I-MIBG therapy. Clin Oncol (R Coll Radiol). 2003 Jun;15(4):193-8. doi: 10.1016/s0936-6555(02)00273-x. PMID 12846498
- [Background] Yadegarfar G, Friend L, Jones L, Plum LM, Ardill J, Taal B, Larsson G, Jeziorski K, Kwekkeboom D, Ramage JK; EORTC Quality of Life Group. Validation of the EORTC QLQ-GINET21 questionnaire for assessing quality of life of patients with gastrointestinal neuroendocrine tumours. Br J Cancer. 2013 Feb 5;108(2):301-10. doi: 10.1038/bjc.2012.560. Epub 2013 Jan 15. PMID 23322194
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Yao JC, Fazio N, Singh S, Buzzoni R, Carnaghi C, Wolin E, Tomasek J, Raderer M, Lahner H, Voi M, Pacaud LB, Rouyrre N, Sachs C, Valle JW, Fave GD, Van Cutsem E, Tesselaar M, Shimada Y, Oh DY, Strosberg J, Kulke MH, Pavel ME; RAD001 in Advanced Neuroendocrine Tumours, Fourth Trial (RADIANT-4) Study Group. Everolimus for the treatment of advanced, non-functional neuroendocrine tumours of the lung or gastrointestinal tract (RADIANT-4): a randomised, placebo-controlled, phase 3 study. Lancet. 2016 Mar 5;387(10022):968-977. doi: 10.1016/S0140-6736(15)00817-X. Epub 2015 Dec 17. PMID 26703889
- See also: EORTC Quality of Life Questionnaire - QLQ-GINET21 — http://qol.eortc.org/questionnaire/qlq-ginet21/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT04831567/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT04831567/ICF_001.pdf